CLINICAL TRIAL: NCT03138720
Title: A Phase II Study of Paclitaxel Protein Bound + Gemcitabine + Cisplatin + Paricalcitol as Pre-operative Treatment in Patients With Untreated Resectable, Borderline Resectable and Locally Advanced Adenocarcinoma of the Pancreas
Brief Title: Pre-operative Treatment for Patients With Untreated Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: HonorHealth Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NABPLAGEM-NEO 2017-001
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Resectable Pancreatic Cancer; Unresectable Pancreatic Cancer; Pancreatic Adenocarcinoma; Neoadjuvant Pancreatic Cancer
MeSH Terms: interventions — Taxes; Albumin-Bound Paclitaxel; Cisplatin; Gemcitabine; paricalcitol

STUDY DESIGN:
Intervention Model Description: There will be two treatment groups: those who are deemed resectable and those that are deemed borderline resectable and with locally advanced pancreas cancer.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental): All patients will receive open label medication at set dosages unless the dosage needs to be adjusted to treat an adverse event or dose toxicity.
  Interventions: Drug: Paclitaxel Protein Bound (Abraxane)

INTERVENTIONS:
Drug: Paclitaxel Protein Bound (Abraxane) — Participants will be treated with the regimen prior to having surgery. Participants will complete 3 cycles (cycle is 21 days) and then will be evaluated for CA19-9 normalization. If CA19-9 is normalized, then participant will be scheduled for surgery and moved to standard of care. If CA19-9 is not normalized then participants will complete another 3 cycles.
  Other Names: Cisplatin (Platinal; Gemcitabine (Gemzar); Paricalcitol (Zemplar)

SUMMARY:
The purpose of this study is to determine if the combination of paclitaxel protein bound, gemcitabine, cisplatin, paricalcitol are effective in individuals with resectable and unresectable pancreatic cancer.

DETAILED DESCRIPTION:
Neoadjuvant therapy has become the consensus treatment for individuals with locally advanced unresectable disease and borderline resectable disease. Typical regimens utilize those that are used in the metastatic setting for pancreatic cancer, such as FOLFIRINOX (5-FU, Leucovorin, Irinotecan, and Oxaliplatin) and paclitaxel protein bound plus Gemcitabine. Currently, the recommendation of utilizing neoadjuvant therapy for potentially resectable pancreatic cancer has been met with controversy. However a recent study published an analysis of individuals with potentially resectable pancreatic cancer and showed a median overall survival of 31.5 months with 44.9 months for the 60 individuals who underwent neoadjuvant therapy and resection compared to 8.1 months for the 9 patients who were not resected. Another study examined the use of nab-paclitaxel, gemcitabine, capecitabine, and cisplatin (PAXG regimen) in individuals with unresectable or borderline resectable pancreatic cancer patients. A partial response was observed in 67% of the patients along with progression-free survival at 6 months being 96%. Furthermore, a recent study examining stage I or stage II pancreas cancer patients who received either neoadjuvant therapy followed by resection or those who received upfront resection was reported. In those receiving neoadjuvant therapy, overall survival was 26 months compared to 21 months. Neoadjuvant, as opposed to adjuvant therapy potentially increases the amount of exposure of drug to the tumor. It allows for the completion of therapy prior to surgery to prevent patient drop-out due to perioperative complication. Neoadjuvant therapy also acts as a selection tool for optimal surgical candidates by identifying aggressive tumor biology prior to surgery and therefore selecting out those who will not benefit from resection. Radiation therapy may be also employed in the neoadjuvant setting as a means to help with local control and survival in individuals without micrometastatic disease.

The combination of nab-paclitaxel (now called paclitaxel protein bound) and gemcitabine had a high response and survival in the phase I and II study in advanced pancreatic cancer. In this phase I study with expansion at the phase II dose, 67 pts were accrued. The phase II dose was determined to be weekly nab-paclitaxel 125 mg/m2 with gemcitabine 1000 mg/m2. Therapy was well tolerated at the phase II dose. For all patients (n=67), the median time for progression-free survival (PFS) was 7.1 months (95%CI, 5.7 to 8.0 months), and the median time for overall survival (OS) was 10.3 months (95% CI, 8.4 to 13.6 months). For patients at the recommended dose of 125 mg/m2 nab-paclitaxel, the median PFS was 7.9 months (95% CI, 5.8 to 11.0 months), and the median OS time was 12.2 months (95% CI, 8.9 to 17.9 months). Additionally, the 1-year survival is reported at 48% at the maximum tolerated dose (MTD), and the overall response rate (ORR) was 46% for all patients (n=67). The combination of nab-paclitaxel and gemcitabine was generally well tolerated and had substantial antitumor activity in patients with pancreatic cancer, enough to warrant a phase III clinical trial.

In the phase III (MPACT study, n=861) patients were randomly assigned to nab-paclitaxel plus gemcitabine (431 patients) or gemcitabine (430). The median overall survival was 8.5 months in the nab-paclitaxel-gemcitabine group as compared with 6.7 months in the gemcitabine group (P<0.001). The one year survival rate was 35% in the nab-paclitaxel-gemcitabine group versus 22% in the gemcitabine group, and 9% versus 4% at 2 years. The median PFS was 5.5 months in the nab-paclitaxel-gemcitabine group, as compared with 3.7 months in the gemcitabine group (P<0.001); the response rate according to independent review was 23% versus 7% in the two groups (P<0.001). Adverse events were tolerable with grade > 3 events of neutropenia (38% in the nab-paclitaxel-gemcitabine group vs. 27% in the gemcitabine group), fatigue (17% vs. 7%), and neuropathy (17% vs. 1%) and febrile neutropenia (3% versus 1%). Based on the results of this study, nab-paclitaxel plus gemcitabine is a FDA approved regimen for pancreatic cancer.

Building on the design and mechanisms of action of the nab-paclitaxel and gemcitabine combination, a prior protocol introduced a third cytotoxic agent cisplatin, was added to this doublet. The rationale for adding cisplatin to nab-paclitaxel and gemcitabine was that in a study of 1,029 patients whose pancreatic cancer tumors were sent for molecular profiling, 57% of these tumors were negative for ERCC1, indicating sensitivity to a platinum anti-tumor agent. In addition to the above, in our whole genome/transcriptome sequencing analysis, we found that abnormal repair pathways were a feature of all of the pancreatic cancers that were sequenced. Cisplatin prevents cellular DNA repair by binding to and causing crosslinking of DNA, triggering apoptosis. Cisplatin has been used in other combination regimens to treat patients with PDA. For example, the cisplatin, epirubicin, 5-fluorouracil and gemcitabine (PEFG) regimen had an acceptable toxicity profile and was associated with a 24% partial response rate, 5 month progression-free survival (PFS) and 8.3 month overall survival as second line therapy.

Prior to 2015, there were no documented reports of the combination of cisplatin with paclitaxel protein bound and gemcitabine in the treatment of any human cancer. However, cisplatin had been combined with paclitaxel and gemcitabine in the treatment of patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) patients and had shown substantial antitumor activity with an acceptable safety profile. In that phase I-II study of 65 patients with advanced NSCLC, the overall response rate was 57%. The aforementioned neoadjuvant study led by Reni also utilized cisplatin with albumin bound paclitaxel along with gemcitabine and capecitabine.

More recently there has been even more compelling science indicating that one should consider DNA repair as an Achilles heel in pancreatic cancer. A team led by Nurse Practitioner Gayle Jameson recently reported on the phase Ib/II trial of the combination of paclitaxel protein-bound plus gemcitabine plus cisplatin. In 24 evaluable patients with stage IV pancreatic cancer they reported a response rate of 71% (Complete Response (CR) + Partial Response (PR)) along with a 88% disease control rate (CR + PR+ Stable Disease (SD) at 9 weeks). Utilizing this highly active therapy in the neoadjuvant setting may lead to further improvement in overall survival and progression free survival in patients with pancreatic cancer.

Most recently the spectacular work of researchers has awakened the world of pancreatic cancer research to the possibility that Vitamin D could be a substantial player in normalizing the tumor microenvironment from an immunologically friendly (to the tumor) one to an immunologically hostile one (e.g. decreased IL6, decreased CXCL12 etc.). In addition, the vitamin D analog decreased production of collagen, decreased Myeloid Derived Suppressor cells (MDSCs) and decreased regulating T cells. In an ongoing neoadjuvant trial utilizing gemcitabine and paclitaxel protein bound with paricalcitol compared to gemcitabine and paclitaxel protein bound, a modulation of the tumor microenvironment has been seen including greater infiltration of CD3 positive lymphocytes. Therefore, a trial utilizing gemcitabine, paclitaxel protein bound, cisplatin and paricalcitol may yield promising results in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically or cytologically confirmed resectable, borderline resectable, or locally advanced (unresectable) PDAC (based upon Tempero et al 2016)

   * Definition of Resectable Pancreatic Cancer includes all of the following:
   * No evidence of extra pancreatic disease
   * No evidence of tumor-arterial abutment (celiac, SMA [superior mesenteric artery] or HA [hepatic artery])
   * If tumor induced narrowing of the SMV [superior mesenteric vein], PV [portal vein] or SMV-PV [superior mesenteric-portal vein] confluence is present, it must be <50% of the diameter of the vessel
   * Definition of Borderline Resectable Pancreatic Cancer
   * To include at least one of the following:
   * Tumor abutment <180° of the SMA or celiac axis
   * Tumor abutment or encasement of a short segment of the HA
   * Tumor induced narrowing of SMV, PV or SMV-PV of >50% of the diameter of the vessel.
   * Short segment occlusion of the SMV, PV or SMV-PV with a suitable PV above and SMV below, for reconstruction
   * Biopsy proven N1 disease (regional lymph nodes involved) from pre-referral biopsy or EUS-guided FNA
   * Definition of Locally Advanced (Unresectable)
   * Artery: Tumor encasement (> 180°) of SMA or celiac artery
   * Vein Occlusion of SMV, PV or SMV-PV without suitable vessels above and below the tumor to allow for reconstruction (no distal or proximal target for vascular reconstruction)
   * No extra pancreatic disease: No evidence of peritoneal, hepatic, or extra-abdominal metastases
2. Age ≥ 18 years.
3. If a female patient is of child-bearing potential, she must have a negative serum pregnancy test (≥β-hCG) documented within 72 hours of the first administration of study drug
4. If sexually active, the patient and partner must agree to use contraception considered adequate and appropriate by the Investigator
5. Patient must have received no prior chemotherapy or radiation therapy for PDAC
6. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count ≥ 1,500/mm3
   * platelets ≥ 100,000/mm3
   * Hematocrit level > 27%
   * total bilirubin within institutional upper limit of normal (ULN)
   * AST/ALT ≤ 2.5 × institutional ULN
   * Alkaline phosphatase (AP) ≤ 2.5 x institutional ULN
   * Creatinine < 1.5 mg/dl
7. Patient has acceptable coagulation status as indicated by an INR ≤ 1.5 x ULN. Patients on anticoagulation can be included at the discretion of the investigator.
8. Karnofsky Performance Status (KPS) of ≥70%.
9. Have an elevated CA 19-9

Exclusion Criteria:

1. Patient will be excluded from this study if any of the following criteria apply: Evidence of metastatic disease. No metastatic disease defined as any one or more of the following:

   * Suspicious lymphadenopathy outside of the standard surgical field (i.e. aortocaval nodes, distant abdominal nodes)
   * Radiographic evidence for metastatic disease in distant organs, peritoneum, or ascites
2. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
3. Known infection with HIV, hepatitis B, or hepatitis C.
4. Has undergone major surgery, other than diagnostic surgery (i.e. surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
5. History of allergy or hypersensitivity to the study drugs.
6. Serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the patient to receive an experimental research drug.
7. Current, serious, clinically significant cardiac arrhythmias as determined by the investigator.
8. Patient is unwilling or unable to comply with study procedures.
9. Patient is enrolled in any other therapeutic clinical protocol or investigational trial.
10. Patient with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
11. Use of non-FDA approved cannabinoids are prohibited. Total daily usage of up to 40 mg per day of marinol is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
CA19-9 value | approximately 63 days
  Laboratory testing will be used to determine if the CA19-9 value has normalized after 3 cycles of treatment.

SECONDARY OUTCOMES:
Pathologic Complete Response Rate | approximately 63 days
  Participants will have an MRI completed after 3 cycles to determine if the tumor has responded to treatment. RECIST 1.1 criteria will be used to evaluate response. A confirmatory PET scan may be ordered to confirm complete response.
Overall Survival | every 12 weeks after study completion
  Participants will be contacted by telephone every 12 weeks until date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Erkut Borazanci, MD, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with outside researchers.